CLINICAL TRIAL: NCT06329973
Title: A Single-arm, Open-label, Multicenter, Phase Ib/II Study to Evaluate the Safety and Efficacy of Fruquintinib in Combination With Sintilimab and CAPEOX as 1L Treatment for Advanced Unresectable or Metastatic G/GEJ Cancer (FUNCTION Research)
Brief Title: Fruquintinib in Combination With Sintilimab and CAPEOX as First-line Treatment for G/GEJ Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-237
Record Dates: First submitted 2024-01-24; First posted 2024-03-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib in combination with Sintilimab and CAPEOX (Experimental)
  Interventions: Drug: Fruquintinib in combination with Sintilimab and CAPEOX

INTERVENTIONS:
Drug: Fruquintinib in combination with Sintilimab and CAPEOX — Different doses of fruquintinib combined with sintilimab and CAPEOX

SUMMARY:
Based on the current status and progress in the treatment of gastric cancer, our center prospectively designed a first-line comprehensive treatment plan for unresectable or postoperative recurrent advanced gastric/gastroesophageal conjoint adenocarcinoma, fruquintinib + sintilimab + oxaliplatin + Capecitabine (CAPEOX), which utilizes the tumor immunomodulation and vascular normalization effects of fruquintinib. While improving the effective perfusion of intravenous chemotherapy with CAPEOX regimen, further combining with PD-1 monoclonal antibody to regulate the immunosuppressive microenvironment and reactivate the anti-tumor immune response of the body. An exploratory dose-climbing trial was designed to evaluate the clinical efficacy and safety of fruquintinib in combination with Sintilimab and CAPEOX in clinical practice. At the same time, changes in genome, pathology and immune microenvironment of tumor-related tissues before and after treatment were observed, and molecular markers related to curative effect were screened to explore the molecular mechanism affecting the curative effect of combination therapy, and further enrichment of therapeutic advantage groups to improve the surgical conversion rate laid the foundation for future large-scale clinical studies

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-75 years (including 18 and 75 years);
2. Understand the research procedure and content, and voluntarily sign a written informed consent;
3. Incurable advanced/recurrent gastric or gastroesophageal junction adenocarcinoma with histopathological and/or cytological confirmation of HER2-negative or HER2 status unknown;
4. There is at least one measurable lesion according to RECIST 1.1 criteria;
5. No previous treatment with VEGFR-targeting drugs or PD-1/PD-L1 monoclonal antibody. Patients who had received platinum or paclitaxel or fluorouracil adjuvant chemotherapy after surgery and recurred more than 6 months after the end of chemotherapy without grade 2 toxicity or higher could be enrolled.
6. Physical condition score (ECOG PS score) : 0-1 score;
7. Expected survival ≥3 months;
8. The main organs function well;That is, the relevant check indicators within 14 days before randomization meet the following requirements:

   Hemoglobin ≥ 90 g/L (no transfusion within 14 days); Neutrophil count > 1.5×109/L; Platelet count ≥ 100×109/L; Total bilirubin ≤ 1.5×ULN (upper limit of normal); Serum glutamic pyruvic aminotransferase (ALT) or serum glutamic oxalacetic aminotransferase (AST) ≤ 2.5×ULN; If there is liver metastasis, ALT or AST ≤ 5×ULN; Endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); Cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%; Thyroid function index: thyroid stimulating hormone (TSH), free thyroxine (FT3/FT4) in the normal range;
9. Weight of more than 40 kg (including 40 kg), or BMI > 18.5
10. Women who are fertile must have a negative urine or serum pregnancy test within 7 days prior to randomization and must consent to use highly effective contraception during the study period and for at least 120 days after the last administration of fruquintinib and sintilimab and for at least 180 days after the last administration of chemotherapy (Appendix 9);
11. Men who are not sterilized must consent to use highly effective contraception during the study period and for at least 120 days after the last administration of fruquintinib and sintilimab and for at least 180 days after the last administration of chemotherapy (Appendix 9).

Exclusion Criteria:

1. Patients with other malignant tumors in the past or at the same time, but have been cured of early tumors, including skin basal cell carcinoma, cervical carcinoma in situ, stage I lung cancer, stage I colorectal cancer and other tumors that researchers judge will not affect the patient's life in the short term can be excluded;
2. Participated in other drug clinical trials within four weeks;
3. have multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction);
4. Have a history of bleeding, any bleeding event with a severity rating of CTCAE5.0 or higher occurring within 4 weeks prior to screening;
5. Patients with known central nervous system metastasis or history of central nervous system metastasis before screening. For patients with clinically suspected CNS metastasis, CT or MRI examination must be performed within 28 days before enrollment to rule out CNS metastasis.
6. Patients with hypertension who are not well controlled by single antihypertensive medication (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90mmHg); Patients with history of unstable angina pectoris; Patients with newly diagnosed angina pectoris or myocardial infarction within 3 months prior to screening; Arrhythmias (including QTcF: ≥450 ms in men and ≥470 ms in women) requiring long-term use of antiarrhythmic drugs and New York Heart Association grade ≥II cardiac insufficiency;
7. long-term unhealed wounds or incomplete healing fractures;
8. Imaging shows that the tumor has invaded important blood vessels, or the investigator determines that the patient's tumor is highly likely to invade important blood vessels during treatment and cause fatal massive bleeding;
9. Patients with abnormal coagulation function and bleeding tendency (14 days before randomization must meet: INR in the normal range without the use of anticoagulants, or no clinically significant abnormalities); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogs; Low doses of warfarin (1 mg orally, once daily) or low doses of aspirin (up to 100 mg daily) are permitted for prophylactic purposes if INR ≤ 1.5;
10. Occurrence of arteriovenous thrombosis events within 6 months prior to screening, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis (except venous thrombosis caused by intravenous catheterization in previous chemotherapy and cured by investigators), pulmonary embolism, etc.;
11. Urine routine indicated urinary protein ≥++ and confirmed 24-hour urinary protein quantity > 1.0g;
12. Have used immunotargeted therapy drugs;
13. Have a history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
14. Patients with infectious pneumonia, non-infectious pneumonia, interstitial pneumonia and other patients requiring corticosteroids;
15. A history of serious chronic autoimmune diseases, such as systemic lupus erythematosus; History of ulcerative enteritis, Crohn's disease and other inflammatory bowel diseases, irritable bowel syndrome and other chronic diarrheal diseases; A history of sarcoidosis or tuberculosis; History of active hepatitis B, hepatitis C and HIV infection; Well controlled non-severe immune diseases such as dermatitis, arthritis, psoriasis, etc. can be included. Hepatitis B virus drops <1000copy/ml could be included in the group.
16. Patients with hypersensitivity to human or murine monoclonal antibodies;
17. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
18. pleural effusion or abdominal effusion with clinical symptoms requiring clinical intervention;
19. Patients who do not follow medical advice, do not use drugs according to regulations, or have incomplete data that can affect the evaluation of efficacy or safety;
20. In the judgment of the investigator, there is a serious concomitant disease that endangers the patient's safety or interferes with the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of enrollment until the date of the end of the study, assessed up to 48 months
  It refers to the proportion of patients whose tumors have shrunk to a certain extent for a certain period of time, including CR and PR cases
Maximum tolerated dose | Within the first 21 days of treatment
  Refers to the maximum tolerated dose of the whole group

SECONDARY OUTCOMES:
Overall Survival | From date of enrollment until the date of death, assessed up to 48 months
  Refers to the date from admission to death from any cause
Progression Free Survival | From date of enrollment until the date of first documented progression, assessed up to 48 months
  Refers to the date from admission to the first onset of disease progression or death from any cause, whichever comes first
Disease Control Rate | From date of enrollment until the date of the end of the study, assessed up to 48 months
  Refers to the percentage of confirmed complete response, partial response, and stable disease cases in patients evaluated for efficacy
Duration of Response | From date of enrollment until the date of the end of the study, assessed up to 48 months
  Refers to the date of first documented response (Complete Response or Partial Response) until the date of first documented disease progression or death from any cause, whichever occurs first.
Surgical conversion rate | From date of enrollment until the date of the end of the study, assessed up to 48 months
  Refers to the proportion of patients with initially unresectable disease who achieve R0/R1 resection after therapy
Adverse events | From first dose of study drug to 30 days after last dose or the initiation of a new anticancer therapy, whichever occurred first, up to the end of study.
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0
Identification of molecular biomarkers predictive of efficacy | From date of enrollment until the date of the end of the study, assessed up to 48 months
  To investigate associations between baseline and on-treatment molecular biomarkers (e.g., expression of PD-L1 and Claudin 18.2, EBEV, MMR, and other factors) with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Chen, Study Chair — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared for secondary analysis under controlled access.
Supporting Information: CSR
Time Frame: Clinical study report will be available within 6 months after article publication on Vivli.
Access Criteria: Proposals require approval by an independent review committee and a signed data use agreement. Access criteria: (1) Meta-analysis of outcomes; (2) Validation of novel biomarkers.
URL: https://clinicaltrials.gov/study/NCT06329973#study-plan

REFERENCES:
- [Derived] Chen B, Zhao J, Lv H, Xu W, Wang J, Nie C, He Y, Zhang B, Huang J, Liu Y, Ma F, Zhang H, Guo Y, Liu Y, Li P, Chen X, Chen X. Single-arm, open-label, multicentre phase 1b/2 study to evaluate the safety and efficacy of fruquintinib combined with sintilimab and CAPEOX as a first-line treatment for advanced gastric or gastroesophageal junction adenocarcinoma (FUNCTION study): a study protocol. BMJ Open. 2025 Sep 26;15(9):e100241. doi: 10.1136/bmjopen-2025-100241. PMID 41005780